CLINICAL TRIAL: NCT07019116
Title: Efficacy of an Artificial Intelligence Algorithm for Gatekeeping in Referrals From Primary Care to Specialized Care: a Randomized Controlled Trial
Brief Title: Efficacy of Artificial Intelligence for Gatekeeping in Referrals to Specialized Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Rio Grande do Sul State Health Department - SES/RS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-0589
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Primary Care; Primary Care Patients With Chronic Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard gatekeeping process (Active Comparator): In standard gatekeeping, the current process will be used without interventions.
  Interventions: Other: Standard gatekeeping; Other: Subsequent interactions between primary care and regulation system
- Artificial Intelligence for Gatekeeping (Experimental): An AI algorithm will perform the first evaluation (triaging) of the referral.
  Interventions: Other: AI algorithm; Other: Subsequent interactions between primary care and regulation system

INTERVENTIONS:
Other: Standard gatekeeping — Human evaluators (mostly physicians) review referrals and determine, based on established protocols, whether they should be authorized.
  Arms: Standard gatekeeping process
Other: AI algorithm — An AI algorithm was developed to perform the first evaluation (triaging) of the referrals inserted in the electronic referral system from the Rio Grande do Sul Health Department.
  Arms: Artificial Intelligence for Gatekeeping
Other: Subsequent interactions between primary care and regulation system — After the first evaluation of a referral, several subsequent rounds of interaction between gatekeepers and primary care physicians can be conducted to further detail patient needs and urgency.

SUMMARY:
In Rio Grande do Sul, Brazil, the demand for specialty care referrals has increased sharply with the adoption of the electronic regulatory system, especially in rural areas. In 2023 alone, over 79,000 referrals were submitted monthly, totaling 1.7 million annual gatekeeping decisions. Due to workforce limitations, nearly 70% of referrals are authorized automatically, often without clinical validation. This leads to delays for high-risk patients, unnecessary specialist visits, and a growing backlog, currently over 172,000 pending referrals. To address this, an AI algorithm was developed to triage referrals based on urgency and appropriateness.

The investigators propose a prospective controlled study with randomized implementation of the AI tool across selected specialty queues in the electronic referral system. The population will consist of referrals from specialties waitlists from municipalities in Rio Grande do Sul. Specialties to be included will be selected by the State Health Department prospectively according to gatekeeping needs. The intervention will be an AI-based triage algorithm. The control will be a standard gatekeeping process. The primary outcome is the proportion of referrals with a final decision (authorized or redirected to primary care) within six months; secondary outcomes include time to decision and appointment, system-level performance metrics. Referrals will be randomly assigned to algorithmic or human gatekeeping with a 1:1 ratio. The algorithm classifies referrals into two groups: not authorized (pending more data or teleconsultation), authorized. Authorization cases are further divided into routine and high-risk referrals to help the manage demand. Each AI prediction provides a probability from 0 to 1 of authorization (or deferring). The implementation threshold is set at 0.8; cases below this level will be classified as low confidence for decision and will not be included. According to the State Health Department's decisions, several referral lines are expected to be selected for the intervention. A sample size 934 (467 per arm) for each included specialty was calculated to detect a 1.2 relative risk for the primary outcome with 90% power and 5% significance.

ELIGIBILITY:
Inclusion Criteria:

* All referrals from a given specialty (waitlist) will be eligible.
* Specialties will be selected following Rio Grande do Sul Health Department priorities.

Exclusion Criteria:

* Referrals that the AI algorithm can not evaluate. These include referrals with attachments (further information in image or PDF files) and referrals with previous rounds of discussion.
* Referrals in which the algorithm has low confidence in the decision (i.e., informed data lead to a decision with a probability below 80%) will not be included in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 934 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Referrals with final decision | 6 months
  The proportion of referrals with a final decision includes those authorized for specialist care and those redirected to primary care without an in-person specialist consultation.

SECONDARY OUTCOMES:
Time to final decision | 6 months
  Time to final decision (authorization or deferral) for the referral.
Time to consult in high-risk patients | 6 months
  Time to specialist appointment for high-priority (red/orange) cases.
Use of remote consultations | 6 months
  Rio Grande do Sul has a provider-to-provider consultation service. The proportion of referrals that used this service will be assessed.
Waitlist size over time | 6 months
  The overall size of the referral waitlist will be assessed before and after the implementation of the algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris V. Rados, Ph.D., Principal Investigator — TelessaúdeRS

IPD SHARING:
Plan to Share IPD: Undecided
Final data responsibility lies with the Rio Grande do Sul State Health Department, and the data are classified as high-risk health data under the Brazilian General Data Protection Law.